CLINICAL TRIAL: NCT07290387
Title: Tele-Savvy for Latino Caregivers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Maria Quinones, Assistant Professor of Clinical Nursing, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00009037; 5P30AG064200 (NIH)
Record Dates: First submitted 2025-12-15; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer Disease; Dementia; Caregiver Stress
MeSH Terms: conditions — Alzheimer Disease; Dementia; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: This is a single arm Stage 1b behavioral clinical trial using a pre post design. All enrolled participants receive the Tele Savvy for Latino Caregivers intervention and outcomes are assessed at baseline immediately post intervention and three months post intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Behavioral: Tele Savvy for Latino Caregivers

INTERVENTIONS:
Behavioral: Tele Savvy for Latino Caregivers — Tele Savvy for Latino Caregivers is a culturally adapted seven week caregiver education and support program delivered remotely. Participants attend weekly ninety minute group sessions via videoconference and receive two to three asynchronous instructional videos per week. The intervention focuses on developing caregiver mastery skills including caregiving competence confidence and stress management.

SUMMARY:
Latino caregivers of individuals with Alzheimer's disease and related dementias experience high levels of stress burden and depressive symptoms and are underrepresented in caregiver intervention research. Tele Savvy is an evidence based caregiver education program that focuses on developing caregiver mastery skills. This study aims to culturally adapt the Tele Savvy intervention for Latino caregivers and evaluate its preliminary efficacy in a Stage 1b single arm clinical trial. The intervention is delivered remotely and includes weekly group sessions and asynchronous instructional videos. Primary outcomes focus on caregiver mastery with secondary outcomes including stress burden depressive symptoms and self efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Identify as Hispanic or Latino
* Age 18 years or older
* Spanish speaking and able to read and write in Spanish
* Provide at least four hours per week of care to a community dwelling loved one with Alzheimer's disease or related dementias
* Have access to an electronic device and internet
* Willing to participate in study interviews and intervention sessions

Exclusion Criteria:

* Physical or sensory conditions preventing use of a computer tablet or smartphone
* Planning to move the care recipient to an institutional setting within six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-12-21 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Mean Change in Caregiver Mastery Score | Baseline to three months post intervention completion
  Caregiver mastery is measured using two Pearlin Caregivers' Stress subscales: Caregiving Competence and Confidence and Management of Situation. Each subscale consists of four Likert type items. Item responses are scored according to published scoring instructions and summed to produce a total caregiver mastery score for each participant at each assessment time point. The outcome is defined as the mean change in the total caregiver mastery score from baseline to three months post intervention across participants.

SECONDARY OUTCOMES:
Mean Change in Perceived Stress Scale Score | Baseline to Three Months Post Intervention
  Perceived stress is measured using the 10 item Perceived Stress Scale. Each item is scored on a Likert type scale according to standard scoring procedures, with designated items reverse scored. Item scores are summed to generate a total Perceived Stress Scale score for each participant at each assessment time point. The outcome is defined as the mean change in the total Perceived Stress Scale score from baseline to three months post intervention.
Mean Change in Total Zarit Caregiver Burden Scale Score | Baseline to Three Months Post Intervention
  Caregiver burden is measured using the Zarit Caregiver Burden Scale. Individual item responses are scored and summed to produce a total Zarit Burden score for each participant at each assessment time point. The outcome is defined as the mean change in the total Zarit Caregiver Burden Scale score from baseline to three months post intervention.
Mean Change in Total CES D R Depression Score | Baseline to Three Months Post Intervention
  Depressive symptoms are measured using the Center for Epidemiologic Studies Depression Scale Revised. Item responses are scored according to standard scoring procedures and summed to generate a total CES D R score for each participant at each assessment time point. The outcome is defined as the mean change in the total CES D R score from baseline to three months post intervention.
Mean Change in Total Family Caregiver Self Efficacy for Managing Dementia Score | Baseline to Three Months Post Intervention
  Caregiver self efficacy is measured using the Family Caregiver Self Efficacy for Managing Dementia questionnaire. Item responses are scored and summed to generate a total self efficacy score for each participant at each assessment time point. The outcome is defined as the mean change in the total caregiver self efficacy score from baseline to three months post intervention.
Mean Total Satisfaction Questionnaire Score Immediately Post Intervention | Immediately following completion of the seven week intervention
  Participant satisfaction is measured using a satisfaction questionnaire administered immediately after intervention completion. Item responses are scored and summed to produce a total satisfaction score for each participant. The outcome is defined as the mean total satisfaction questionnaire score across participants.

IPD SHARING:
Plan to Share IPD: No